CLINICAL TRIAL: NCT05721846
Title: Phase 1 Study of Nivolumab With Ipilimumab Combined With TGFβ-15 Peptide Vaccine and Stereotactic Body Radiotherapy for Refractory Pancreatic Cancer (CheckVAC)
Brief Title: Nivolumab With Ipilimumab Combined With TGFβ-15 Peptide Vaccine and Radiotherapy for Pancreatic Cancer
Acronym: CheckVAC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inna Chen, MD (Other)
Responsible Party: Sponsor-Investigator, Inna Chen, MD, Lead of the Pancreatic Cancer Center, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA 2217
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): SBRT: 15 Gy x 1 on a single site of disease on day 1 cycle 1
  Immunotherapy:
  Nivolumab 3 mg/kg (up to 240 mg maximum) as i.v. infusion on day 1 (± 3 days) of each 14-day treatment cycle Ipilimumab 1 mg/kg as i.v. infusion on day 1 cycle 1 and subsequently every 6 weeks (± 3 days).
  Vaccine (500 μl aqueous solution of 200 μg TGFβ-B-15 peptide mixed to an emulsion with 500μl Montanide ISA-51) as s.c. injection on day 1 of the first 6 cycles and subsequently every 4 weeks (± 3 days)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Radiation: SBRT; Biological: TGFβ-B-15 peptide

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg (up to 240 mg maximum) as i.v. infusion on day 1 (± 3 days) of each 14-day treatment cycle
Drug: Ipilimumab — 1 mg/kg as i.v. infusion on day 1 cycle 1 and subsequently every 6 weeks (± 3 days)
Radiation: SBRT — SBRT: 15 Gy x 1 on a single site of disease on day 1 cycle 1
Biological: TGFβ-B-15 peptide — Vaccine (500 μl aqueous solution of 200 μg TGFβ-B-15 peptide mixed to an emulsion with 500μl Montanide ISA-51) as s.c. injection on day 1 of the first 6 cycles and subsequently every 4 weeks (± 3 days)

SUMMARY:
"Non-immunogenicity" of PC with high prevalence of immunosuppressive cells and typically a scarcity of tumor-infiltrating effector lymphocytes is considered as one of the reasons for lacking responsiveness to single-agent immunotherapies. Considering the emerging role of the tumor microenvironment, the combination of checkpoint blocking antibodies with immunomodulation of the tumor microenvironment could lead to better responses in tumor historically resistant to radiation and checkpoint blocking antibody approaches as single modalities. For example, the data from the phase 2 study CheckPAC (NCT02866383) showed durable clinical benefit in a small subgroup of patients after adding SBRT of 15 Gy to a combination of nivolumab and ipilimumab (presented at ASCO GI 2022, San Fransisco) in patients with resistant metastatic PC. Furthermore, we have found that the TGFβ-15 immune response is corelated to clinical benefit, supporting the rationale for combining of TGFβ-15 peptide vaccine with CheckPAC strategy (SBRT of 15 in combination with nivolumab and ipilimumab).

DETAILED DESCRIPTION:
SBRT: 15 Gy x 1 on a single site of disease on day 1 cycle 1

Immunotherapy:

Nivolumab 3 mg/kg (up to 240 mg maximum) as i.v. infusion on day 1 (± 3 days) of each 14-day treatment cycle Ipilimumab 1 mg/kg as i.v. infusion on day 1 cycle 1 and subsequently every 6 weeks (± 3 days).

Vaccine (500 μl aqueous solution of 200 μg TGFβ-B-15 peptide mixed to an emulsion with 500μl Montanide ISA-51) as s.c. injection on day 1 of the first 6 cycles and subsequently every 4 weeks (± 3 days)

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histological or cytological confirmation of advanced pancreatic carcinoma prior to entering this study
* Prior therapy requirements:

  * There is no upper limit on the number of prior chemotherapy regimens received. Participants must have received and progressed during or after at least 1 line of systemic chemotherapy in the metastatic setting (gemcitabine or 5-FU based regimens).
  * Notes:

    * If a participant received adjuvant/neoadjuvant systemic combinational therapy, and progressed within 6 months, the adjuvant/neoadjuvant treatment will be considered as 1 line of systemic treatment.
    * In general, discontinuation of 1 drug in a multi-drug regimen and continuation of other drug(s), is considered part of the same line of treatment. Restarting the same regimen after a drug holiday or maintenance chemotherapy can also be considered part of the same line of treatment. Switching from IV (5-FU) to an oral formulation (capecitabine) of the same drug is also considered part of the same line of treatment
    * Minimum time from first systemic therapy for recurrent/metastatic adenocarcinoma of pancreas to progression should be at least 3 months
* Age 18 years and older
* ECOG Performance Status (PS) 0-1
* All participants will be required to undergo mandatory pre- and on-treatment biopsies at acceptable clinical risk as judged by the investigator. An archival pre-treatment sample is not acceptable.
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
  * Platelet count ≥ 75 x 10⁹/L
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * AST/ALT ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of childbearing potential (WOCBP) must use method(s) of contraception as indicated in Appendix 3. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. WOCBP should therefore use an adequate method to avoid pregnancy during the treatment and for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus thetime required for the investigational drug to undergo five half-lives. The half-life of nivolumab is up to 25 days. Men who are sexually active with WOCBP must continue contraception during the treatment and for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Subjects must have signed and dated a BIOPAC approved written informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Participants with active, known or suspected autoimmune disease. Participants are permitted to enroll with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of nivolumab, ipilimumab and radiation in combination with TGFβ-15 peptide vaccine. The following are exceptions to this criterion:

  * Intranasal, inhaled, or topical steroids; or local steroid injections (e.g. intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
* Participants should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and Adverse Drug Reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* WOCBP who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 6 months

SECONDARY OUTCOMES:
Overall response rate | 12 months
Overall survival | 12 months
Progression free survival | 6 months
Duration of response | 12 months
Best overall response | 6 months
Disease control rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No